CLINICAL TRIAL: NCT02505906
Title: Late Toxicity in Breast Cancer Patients Treated With Breast-conserving Surgical Procedures and Radiotherapy Using the Simultaneous Integrated Boost Technique
Acronym: FUSIB
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: SFP2008-06
Record Dates: First submitted 2015-07-15; First posted 2015-07-22 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Late toxicity; Simultaneous integrated boost (SIB); Radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Simultaneous Integrated Boost Technique

SUMMARY:
In summary, breast conserving therapy (BCT) is an effective, save and widely used treatment technique for early breast cancer. Radiotherapy has shown to give better local control and survival benefit and is an integrated part of BCT. The simultaneous integrated boost (SIB) technique is a new treatment technique in breast irradiation. In this technique the whole breast is irradiated simultaneous with boosting the tumour bed, as part of BCT. Late radiation-induced toxicity has not been investigated in patients treated with radiotherapy using this technique. Proposed study will study the late radiation-induced toxicity, describe patients-rated complaints, quality of life, survival and local control curves in patients treated for early breast cancer with breast-conserving surgery in combination with radiotherapy with the SIB technique as compared to sequential radiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* WHO performance status 0-2.
* Invasive breast cancer or ductal carcinoma in situ (DCIS).
* Stage I-III breast cancer or DCIS.
* Treated with curative radiotherapy of the breast (as part of breast conserving therapy) with simultaneous integrated boost technique, with or without irradiation of the regional (including internal mammary) lymph nodes.

Exclusion Criteria:

* Previous thoracic radiotherapy.
* Previous history of malignancy, except adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin.
* Bilateral (synchrone) invasive breast cancer.
* Treatment prior to surgery (i.e. neoadjuvant chemotherapy, neoadjuvant hormonal therapy, pre-operative radiotherapy).
* Distant metastases at diagnosis (M1).
* Unsufficient knowledge of Dutch language.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer treated with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 5043 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Late radiation-induced toxicity (grade 2 or higher) | At 1 year after completion of radiation therapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)
Late radiation-induced toxicity (grade 2 or higher) | At 2 years after completion of radiation therapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)
Late radiation-induced toxicity (grade 2 or higher) | At 3 years after completion of radiation therapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)
Late radiation-induced toxicity (grade 2 or higher) | At 4 years after completion of radiation therapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)
Late radiation-induced toxicity (grade 2 or higher) | At 5 years after completion of radiation therapy
  Toxicity score using Common Terminology for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Overall survival | At 1,2,3,4 and 5 years after completion of radiation therapy
Patient-rated symptoms | At 1,2,3,4 and 5 years after completion of radiation therapy
  Questionnaire: BCSCQ
Quality of life in breast cancer patients treated with radiotherapy after breast conserving surgery | At 1,2,3,4 and 5 years after completion of radiation therapy
  Questionnaires: European Organization for Research and Treatment of Cancer Quality of Life - Core Questionnaire (EORTC QLQ-C30), Quality of Life Questionnaire - Breast Cancer Module (QLQ-BR23) and Adult Comorbidity Evaluation (ACE-27)
Recurrence (local) | At 1,2,3,4 and 5 years after completion of radiation therapy
  Assessed by Mammography, MRI (optional). If indicated: chest X-ray, bone scan, ultrasound
Recurrence (regional) | At 1,2,3,4 and 5 years after completion of radiation therapy
  Assessed by Mammography, MRI (optional). If indicated: chest X-ray, bone scan, ultrasound
Recurrence (distant metastasis) | At 1,2,3,4 and 5 years after completion of radiation therapy
  Assessed by Mammography, MRI (optional). If indicated: chest X-ray, bone scan, ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands